CLINICAL TRIAL: NCT03590990
Title: Diagnostic Outcomes Of The Females Presenting With Breast Lump In Surgical
Brief Title: Diagnostic Outcomes Of The Females Presenting With Breast Lump In Surgical Department Services Hospital Lahore
Status: Completed | Type: Observational
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr. SamiUllah, Medical Officer, Services Hospital, Lahore
Other Study IDs: shabbar246
Record Dates: First submitted 2018-07-07; First posted 2018-07-18 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Breast Lump in Females Presenting to Surgical OPD
MeSH Terms: interventions — Mammography; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasonsography, mammography, biopsy — Ultrasonsography of lump in breast Mammography of patents above 35 years Biopsy if indicated

SUMMARY:
It is a simple crossectional study in which we are trying to identify the outcomes of female breast lump presenting to surgical OPD of services hospital lahore.

ELIGIBILITY:
Inclusion Criteria:female patients with breast lump aged from 20 to onwards

-

Exclusion Criteria:

* female patients with breast abscess

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Study Population: population from lahore with adjacent towns
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Outcome of breast lump in female patients | 4 weeks
  Outcome will either benign disease like fibroadenoma or malignat like carcinoma

IPD SHARING:
Plan to Share IPD: Undecided